CLINICAL TRIAL: NCT05308563
Title: Fall Risk Assessment Using Hybrid Machine Learning and Deep Learning Approaches and a Novel Posturography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other); National Yunlin University of Science and Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202112114RINA
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Age Problem; Fall
Keywords: fall risk; posturography; machine learning; fall efficacy; deep learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Trunk displacement trajectories recorded by the posturography
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this project is to combine a novel posturogrpahy based on HTC VIVE trackers and hybrid machine learning and deep learning algorithms to establish a set of simple, convenient and valid fall risk assessment tool. This observational and follow up study will community elderly aged over 60 years old. The investigators will collect demographic data, questionnaire surveys, traditional balance tests and the tracker-based posturography to obtain the trunk stability parameters in different standing task. The fall risk will be classified according to self-reported falls n the past one year and verified in a 6-month follow up. The investigators will evaluate the performance of different hybrid machine learning and deep learning algorithm to extract the important features of multiple posturographic parameters and select an optimal model. The investigators will use the receiver operating characteristic curve analysis to compute the sensitivity, specificity and accuracy of different algorithms for risk classification and also compare the performance with traditional balance assessment tools.

DETAILED DESCRIPTION:
The purpose of this project is to combine a novel posturogrpahy based on HTC VIVE trackers and hybrid machine learning and deep learning algorithms to establish a set of simple, convenient and valid fall risk assessment tool. This observational and follow up study will community elderly aged over 60 years old. The investigators will collect demographic data, questionnaire surveys, traditional balance tests (Berg Balance scale, Timed-up-and-go, 30s-sit-to-stand, four-stage balance tests) and a tracker-based posturography to obtain the trunk stability parameters in different standing task. The fall risk will be classified according to self-reported falls in the past one year and verified in a 6-month follow up.

The investigators will evaluate the performance of different hybrid machine learning and deep learning algorithm to extract the important features of multiple posturographic parameters and select an optimal model. The investigators will use the receiver operating characteristic curve analysis to compute the sensitivity, specificity and accuracy of different algorithms for risk classification and also compare the performance with traditional balance assessment tools. The investigators will evaluate the correlation of these posturographic features and data obtained by other methods. Risk factors of previous falls and future falls will also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* can walk in the household without device independently

Exclusion Criteria:

* with terminal disease
* with cognitive impairment to follow verbal instruction
* with neurological conditions that are associated with leg weakness
* with significant visual impairment that interferes with daily living and walking

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-living aged group
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of fall events | 6 months
  self-reported fall events according to a followup questionnaire and defined as the sudden, involuntary transfer of body to the ground and at a lower level than the previous one

REFERENCES:
- [Background] Liang HW, Chi SY, Chen BY, Hwang YH. Reliability and Validity of a Virtual Reality-Based System for Evaluating Postural Stability. IEEE Trans Neural Syst Rehabil Eng. 2021;29:85-91. doi: 10.1109/TNSRE.2020.3034876. Epub 2021 Feb 25. PMID 33125332